CLINICAL TRIAL: NCT03656744
Title: A Proof-of-Concept and Dose-Ranging Study Investigating the Efficacy and Safety of HTD1801 in Adults With NASH and T2DM
Brief Title: A Study of HTD1801 in Adults With Nonalcoholic Steatohepatitis (NASH) and Type 2 Diabetes Mellitus (T2DM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: HighTide Biopharma Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HTD1801.PCT012
Record Dates: First submitted 2018-08-30; First posted 2018-09-04 (Actual); Results first posted 2021-12-29 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-11

CONDITIONS: Fatty Liver, Nonalcoholic; NAFLD; Nonalcoholic Fatty Liver Disease; Nonalcoholic Steatohepatitis; Digestive System Diseases; Type 2 Diabetes Mellitus (T2DM)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Digestive System Diseases; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- 500mg HTD1801, bid (Experimental)
  Interventions: Drug: HTD1801
- 1000mg HTD1801, bid (Experimental)
  Interventions: Drug: HTD1801
- placebo, bid (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HTD1801 — HTD1801 tablets, 250mg
  Arms: 1000mg HTD1801, bid; 500mg HTD1801, bid
Drug: Placebo — tablets manufactured to mimic HTD1801 tablets
  Arms: placebo, bid

SUMMARY:
Randomized, double-blind, placebo-controlled, parallel-group study comparing multiple doses of HTD1801 to placebo.

DETAILED DESCRIPTION:
This 18-week randomized, double-blind, parallel-group, proof of concept (POC), dose-ranging study compared multiple doses of HTD1801 to placebo in a 1:1:1 ratio. Since accumulation of hepatic fat is considered the "first hit" in the pathogenesis of NASH (Adams and Angulo 2006), change in liver fat content (LFC) by magnetic resonance imaging estimated proton density fat fraction (MRI-PDFF) is an appropriate primary endpoint and is consistent with that used in other recent Phase 2 POC studies in NASH (Harrison et al., 2018, Madrigal Pharmaceuticals 2018).

The Harrison et al., 2018, Madrigal Pharmaceuticals 2018 study showed clinically meaningful absolute and relative reductions in LFC assessed by MRI-PDFF over 12-week treatment periods thus, it was considered that an 18 week HTD1801 treatment period would therefore be adequate to assess the study's primary endpoint and to maximize collection of exposure and safety related data.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of NASH as assessed by MRI
* Clinically documented diagnosis of T2DM
* Body mass index (BMI) >25 kg/m2

Exclusion Criteria:

* Liver disease unrelated to NASH
* Poorly controlled T2DM or Type 1 Diabetes Mellitus
* History of alcohol or substance abuse or dependence
* Inability to undergo MRI for any reason
* History of significant cardiovascular disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 101 (Actual)
Dates: Start 2018-11-26 (Actual); Primary Completion 2020-02-07 (Actual); Study Completion 2020-03-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Di Bisceglie, MD,FACP,FAASLD, Study Director — HighTide Therapeutics USA, LLC
Locations (17):
- United States (17):
  - Institute for Liver Health, Chandler, Arizona
  - Institute for Liver Health, Tucson, Arizona
  - Adobe Clinical Research, Tucson, Arizona
  - National Research Institute, Panorama City, California
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Florida Research Institute, Lakewood Rch, Florida
  - Compass Research, Orlando, Florida
  - Kansas City Research Institute, Kansas City, Missouri
  - Cumberland Research Associates, Fayetteville, North Carolina
  - Gastro One, Germantown, Tennessee
  - Digestive Health Research, Hermitage, Tennessee
  - Pinnacle Clinical Research, Austin, Texas
  - Doctors Hospital at Renaissance, Edinburg, Texas
  - Pinnacle Clinical Research, San Antonio, Texas
  - Texas Digestive Disease Consultants, Southlake, Texas
  - Harborview Medical Center, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Harrison SA, Gunn N, Neff GW, Kohli A, Liu L, Flyer A, Goldkind L, Di Bisceglie AM. A phase 2, proof of concept, randomised controlled trial of berberine ursodeoxycholate in patients with presumed non-alcoholic steatohepatitis and type 2 diabetes. Nat Commun. 2021 Sep 17;12(1):5503. doi: 10.1038/s41467-021-25701-5. PMID 34535644

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Started | 34 | 34 | 33
Completed | 29 | 27 | 32
Not Completed | 5 | 7 | 1
Not completed — Adverse Event | 1 | 4 | 1
Not completed — Protocol Violation | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Randomized in error. Did not start investigational product. Considered an ET. | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: One-hundred one subjects were randomized into the study, however, subject did not receive investigational study drug and was not included in the efficacy or safety analyses data sets.
Groups:
- Total: Total of all reporting groups
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid | Total
Number analyzed (Participants) | 33 | 34 | 33 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: One subject was randomized in error and did not receive investigational study drug.
  years | 58 (10.2) | 53 (12.2) | 58 (10.7) | 56 (11.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: One subject randomized in error and did not receive investigational study medication.
  Participants
    Female | 26 | 24 | 22 | 72
    Male | 7 | 10 | 11 | 28
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: One subject randomized in error and did not receive investigational study drug.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0
    Asian | 1 | 1 | 0 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
    Black or African American | 3 | 2 | 0 | 5
    White | 29 | 31 | 31 | 91
    More than one race | 0 | 0 | 2 | 2
    Unknown or Not Reported | 0 | 0 | 0 | 0
All Randomized Subjects [Count of Participants; unit: Participants] — Results are reported for all subjects who signed the Institutional Review Board (IRB) approved informed consent form and were randomized into the study. One subject was randomized in error but did not receive investigational study drug and was not included in the analyses efficacy and safety datasets.
  Participants
    Disposition | 33 | 34 | 33 | 100
    Eligible Subjects | 32 | 33 | 33 | 98

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Liver Fat Content (LFC) as Measured by MRI-PDFF
Description: The primary endpoint was the absolute change in liver fat content (LFC) as measured by magnetic resonance imaging derived proton density fat fraction (MRI-PDFF) from Baseline to Week 18.
Time Frame: Baseline through study Week 18
Population: Efficacy set which included all subjects who completed at least 80 days of study drug and had a Week 18 or Early Termination (ET) visit MRI-PDFF assessment.
Measure: Mean (Standard Deviation); unit: Change in percentage of liver fat
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 30 | 27 | 32
Change in percentage of liver fat | -2.918 (4.0204) | -4.829 (4.3516) | -1.962 (4.8844)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.199, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.011, ANCOVA

2. Secondary Outcome: Change in Fasting Glucose
Description: Change in fasting glucose from Baseline to Week 18 .
Time Frame: Baseline through study Week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data available for the change in glucose endpoint.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 26 | 32
mg/dL | 120 (28.6) | 129 (42.5) | 131 (40.9)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.152, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.109, ANCOVA

3. Secondary Outcome: Changes in Hemoglobin A1c
Description: Changes in HbA1c from Baseline to Week 18.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data available for change in hemoglobin A1c endpoint..
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 26 | 32
Percentage | -0.3 (0.68) | -0.6 (0.96) | 0.1 (0.82)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.034, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.004, ANCOVA

4. Secondary Outcome: Proportion of Subjects Who Achieved ≥ 30% Relative Reduction in LFC as Measured by MRI-PDFF
Description: Proportion of subjects who achieved ≥ 30% relative reduction in liver fat content (LFC) as measured by magnetic resonance imaging derived proton density fat fraction (MRI-PDFF) from Baseline to Week 18.
Time Frame: Baseline through study week 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 30 | 27 | 32
Participants | 6 | 10 | 7
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.884, Regression, Logistic
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.236, Regression, Logistic

5. Secondary Outcome: Relative Change in LFC as Measured by MRI-PDFF
Description: Relative change in liver fat content (LFC) as measured by magnetic resonance imaging derived proton density fat fraction (MRI-PDFF) from Baseline to Week 18.
Time Frame: Baseline through study week 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage change
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 30 | 27 | 32
Percentage change | -15.097 (22.7749) | -24.140 (21.7020) | -8.322 (24.4804)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.196, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.016, ANCOVA

6. Secondary Outcome: Number of Subjects Who Normalized LFC to <5% as Measured by MRI-PDFF
Description: Number of subjects who normalized liver fat content (LFC) to <5% as measured by magnetic resonance imaging derived proton density fat fraction (MRI-PDFF) at Week 18.
Time Frame: Baseline through study Week 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 30 | 27 | 32
Participants | 1 | 0 | 0
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.294, Cochran-Mantel-Haenszel

7. Secondary Outcome: Number of Subjects Who Achieved ≥5% Absolute Reduction in Liver Fat Content (LFC) as Measured by MRI-PDFF
Description: Number of subjects who achieved ≥5% absolute reduction in liver fat content (LFC) as measured by magnetic resonance imaging derived proton density fat fraction (MRI-PDFF) from Baseline to Week 18.
Time Frame: Baseline through study Week 18
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 30 | 27 | 32
Participants | 10 | 12 | 8
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.287, Regression, Logistic
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.090, Regression, Logistic

8. Secondary Outcome: Change in HOMA-IR
Description: Change in homeostasis model assessment-estimated insulin resistance (HOMA-IR) from Baseline to Week 18. The higher the HOMA-IR score, the more insulin resistant a person is. Values of <1 are considered optimal while values >2.9 indicate significant insulin resistance.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data was available for the changes in HOMA-IR endpoint and included 4 more subjects than were in the Efficacy set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 26 | 32
score on a scale | -3.38 (6.779) | -4.21 (7.074) | -6.66 (17.752)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.201, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.534, ANCOVA

9. Secondary Outcome: Change in LDL-c
Description: Change in low-density lipoprotein cholesterol (LDL-c) from Baseline to Week 18.
Time Frame: Baseline visit through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data was available for the changes in LDL-c endpoint and included 4 more subjects than were in the Efficacy set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 27 | 25 | 29
mg/dL | 5 (34.1) | -16 (26.5) | 0 (20.5)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.955, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.072, ANCOVA

10. Secondary Outcome: Change in Serum Triglycerides
Description: Change in serum triglycerides from Baseline to Week 18.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited subjects with data was available for the changes in serum triglycerides endpoint and included 4 more subjects than were in the Efficacy set.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 26 | 32
mg/dL | -41 (136.3) | -24 (70.4) | 18 (142.9)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.041, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.120, ANCOVA

11. Secondary Outcome: Change in HDL-c
Description: Change in high-density lipoprotein cholesterol (HDL-c) from Baseline to Week 18.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data was available for the change in HDL-c endpoint and included 4 more subjects than were in the Efficacy set..
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 26 | 32
mg/dL | 1 (5.7) | 0 (8.2) | 0 (7.5)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.955, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.072, ANCOVA

12. Secondary Outcome: Change in AST
Description: Absolute change in aspartate aminotransferase (AST) from Baseline to Week 18.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures included subjects with data was available for the change in AST endpoint and included 4 more subjects than were in the Efficacy set.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 26 | 32
U/L | 0 (13.2) | -13 (26.3) | -3 (11.6)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.488, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.022, ANCOVA

13. Secondary Outcome: Change in ALT
Description: Absolute change in alanine aminotransferase (ALT) from Baseline to Week 18.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data available for the absolute change in alanine aminotransferase endpoint and had 4 more subjects than were in the Efficacy set.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 26 | 32
U/L | -4 (17.9) | -19 (27.2) | -3 (19.2)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.674, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.030, ANCOVA

14. Secondary Outcome: Proportion of Subjects With Elevated ALT at Baseline Who Normalized ALT at Week 18
Description: Proportion of subjects with elevated alanine aminotransferase (ALT) at Baseline who normalized ALT at Week 18.
Time Frame: Baseline through study week 18
Population: Subjects with elevated alanine aminotransferase (ALT) at Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 14 | 18 | 20
Participants | 3 | 9 | 5
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.588, Regression, Logistic
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.103, Regression, Logistic

15. Secondary Outcome: Change in Pro-Peptide of Type III Collagen (Pro-C3)
Description: Change in Pro-C3 from Baseline to Week 18 for subjects with elevated Pro-C3 at Baseline.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data was available for the change in Pro-C3 endpoint and included 4 more subjects than were in the Efficacy set...
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 26 | 32
ng/mL | 0.5 (5.17) | -2.3 (7.09) | -0.8 (2.94)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.236, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.944, ANCOVA

16. Secondary Outcome: Change in ELF Score
Description: Change in the enhanced liver fibrosis (ELF) score. The ELF score is calculated using a published algorithm combining the values of a set of extracellular matrix markers, including TIMP-1, PIIINP, and HA. The ELF score has been reported to show good correlations with fibrosis stages in chronic liver disease, with higher ELF scores associated with higher fibrosis stages. The ELF score is hence used as a prognostic marker for disease progression: ELF score < 9.8 : Low risk of progression, ELF score 9.8 to < 11.3 : Moderate risk of progression and ELF score > = 11.3 : High risk of progression.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data available for the change in ELF score endpoint and include 4 more subjects than were in the Efficacy set.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 25 | 32
score on a scale | 0.05 (0.723) | -0.10 (0.592) | -0.05 (0.461)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.267, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.911, ANCOVA

17. Secondary Outcome: Change in TIMP-1
Description: Change in tissue inhibitor of metalloproteinases 1 (TIMP-1) from Baseline to Week 18.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data available for the change in TIMP-1 endpoint and include 4 more subjects than were in the Efficacy set.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 26 | 32
µg/L | 1.8 (53.26) | -8.9 (57.32) | -6.0 (31.55)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.387, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.855, ANCOVA

18. Secondary Outcome: Change in PIIINP
Description: Change in N-terminal pro-peptide of type III collagen (PIIINP) from Baseline to Week 18.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data available for the change in PIIINP and included 4 more subjects than were in the Efficacy set.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 25 | 32
µg/L | 0.68 (2.905) | 0.03 (3.360) | -0.31 (2.016)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.107, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.489, ANCOVA

19. Secondary Outcome: Change in HA
Description: Change in hyaluronic acid (HA) from Baseline to Week 18.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data available for the change in HA and included set had 4 more subjects than were in the Efficacy set.
Measure: Mean (Standard Deviation); unit: µg/L
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 29 | 25 | 32
µg/L | -0.64 (35.398) | -5.25 (34.046) | -3.83 (49.844)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.515, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.887, ANCOVA

20. Secondary Outcome: Change in Total Bile Acids
Description: Changes in total bile acids from Baseline to Week 18.
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data available for the change in total bile acids and included for 4 more subjects than were in the Efficacy set.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 11 | 12 | 13
μmol/L | 1307 (1432.6) | 1625 (2332.2) | -581 (1487.4)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.003, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.016, ANCOVA

21. Secondary Outcome: Change in FGF19
Description: Change in fibroblast growth factor 19 (FGF19) from Baseline to Week 18
Time Frame: Baseline through study week 18
Population: The Modified Efficacy set was utilized for analyses of secondary endpoints, as well as select analyses of LFC. This analysis set included all randomized subjects who received at least one dose of study drug and who had at least one post-dose MRI-PDFF assessment. The summary measures are additionally limited to those subjects with data available for the change in FGF-19 and include 4 more subjects than were in the Efficacy set.
Measure: Mean (Standard Deviation); unit: μmol/L
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 11 | 12 | 13
μmol/L | -11 (111.8) | -9 (71.1) | -40 (84.8)
Statistical Analysis 1: Comparison: 500mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.124, ANCOVA
Statistical Analysis 2: Comparison: 1000mg HTD1801, Bid vs Placebo, Bid; Test type: Superiority; p = 0.171, ANCOVA

22. Secondary Outcome: Number of Participants Reporting an Adverse Events From Baseline Through Week 18
Description: AEs were mapped to MedDRA version 20.1 preferred term (PT) and system organ class (SOC). If the subject experienced multiple events that mapped to a single preferred term, the greatest severity grade according to CTCAE Version 4.0, and strongest investigator assessment of relation to study medication was assigned to the preferred term. If an event had a missing severity or relationship, it was classified as having the highest severity and/or strongest relationship to study medication. The occurrence of TEAEs was summarized by treatment group by SOC, PT, and severity. Separate summaries of treatment-emergent serious adverse events (SAEs), TEAEs related to study drug, severe or life threatening TEAEs, and TEAEs leading to the discontinuation of study treatment were generated. Additionally, the occurrence of liver-specific AEs was summarized by treatment group. All reported adverse events were listed for individual subjects showing verbatim term, PT and SOC.
Time Frame: Adverse events were collected from the time the subject signed the informed consent form through the date of the last visit for a specific subject, that is, approximately 24 weeks in total for a completed subject.
Population: All subjects included in the safety set.
Measure: Count of Participants; unit: Participants
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
Number analyzed (Participants) | 33 | 34 | 33
Participants | 21 | 26 | 20

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed the informed consent form through the date of the last visit for a specific subject, that is, approximately 24 weeks for a completed subject.
Arm/Group | 500mg HTD1801, Bid | 1000mg HTD1801, Bid | Placebo, Bid
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/34 | 0/33
Serious Adverse Events (participants affected / at risk) | 1/33 | 1/34 | 1/33
Other Adverse Events (participants affected / at risk) | 21/33 | 26/34 | 20/33
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 500mg HTD1801, Bid (N=33) | 1000mg HTD1801, Bid (N=34) | Placebo, Bid (N=33)
Decreased oxygen saturation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Subject was admitted to hospital for elective surgery (left shoulder arthroscopic surgery). Postoperatively, subject developed hypoxia and was placed on oxygen. Hospitalization was prolonged.
Myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) — SAE of MI occurred on Study Day 112 and resolved same day. Presented to emergency with complaint of sharp substernal chest pain. Had severe distal RCA/r PDA disease. Successful per cutaneous intervention performed. Study drug discont. Unrelated.
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Bladder transitional cell carcinoma requiring hospitalization. after presenting to hospital on Study Day 116 with hematuria. Resolved Study Day 117. Unrelated.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 500mg HTD1801, Bid (N=33) | 1000mg HTD1801, Bid (N=34) | Placebo, Bid (N=33)
Infections and Infestations (Infections and infestations) | 4 (4) | 5 (5) | 11 (18) — Upper respiratory tract infection, Nasopharyngitis, bronchitis, gastroenteritis viral,
Gastrointestinal Disorders (Gastrointestinal disorders) | 14 (27) | 19 (40) | 10 (19) — Diarrhea, nausea, abdominal pain upper, abdominal pain, constipation, flatulence, gastroesophageal reflux disease,
Nervous system disorders (Nervous system disorders) | 3 (3) | 5 (6) | 3 (4) — Headache
General Disorders (General disorders) | 2 (5) | 3 (4) | 0 (0) — Fatigue, investigations (alanine aminotransferase increased, blood glucose decreased)
Respiratory disorders (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (2) | 3 (6) — Cough, nasal congestion, sinus congestion
Metabolic disorders (Metabolism and nutrition disorders) | 0 (0) | 2 (4) | 2 (3) — Decreased appetite, dehydration, diabetes mellitus inadequate control, hypertriglyceridemia
Skin disorders (Skin and subcutaneous tissue disorders) | 1 (2) | 2 (3) | 1 (1) — Rash, alopecia
Injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2) — Corneal abrasion, heat exhaustion, joint injury
Endocrine Disorders (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0) — Hypothyroidism,

LIMITATIONS AND CAVEATS:
The study was conducted exclusively in the United States and data may not be applicable to other populations. The study enrolled subjects with presumed NASH and diabetes. Further studies to determine the effect of HTD1801 in non-diabetics may be needed. Future studies will focus on patients with biopsy confirmed NASH and use liver histology (i.e., liver biopsies) as a histological endpoint.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-03-27): https://cdn.clinicaltrials.gov/large-docs/44/NCT03656744/Prot_000.pdf
  • Statistical Analysis Plan (2020-03-25): https://cdn.clinicaltrials.gov/large-docs/44/NCT03656744/SAP_001.pdf